CLINICAL TRIAL: NCT01938118
Title: Mothers and Others: Family-based Obesity Prevention for Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-0510; 1R01HD073237-01 (NIH)
Record Dates: First submitted 2013-08-09; First posted 2013-09-10 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Infant diet; Family diet; Responsive feeding; Infant temperament; Physical activity; Television
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obesity Prevention Group (Experimental): Mothers and families receive a developmentally appropriate educational intervention designed to promote healthy lifestyle behaviors for prevention of excessive weight gain between birth to 15 months of life. Educational content is delivered through eight home visits, five newsletters and twice weekly text messages. At several time points the mother identifies another family member/caregiver to actively participate in the program with her.
  Interventions: Behavioral: Obesity Prevention Group
- Injury Prevention Group (Active Comparator): Mothers and families receive a developmentally appropriate educational intervention designed to promote automobile and home safety behaviors for prevention of childhood injury. Educational content is delivered through eight home visits, five newsletters and twice weekly text messages. At several time points the mother identifies another family member/caregiver, who is only asked to complete surveys/assessments.
  Interventions: Behavioral: Injury Prevention Group

INTERVENTIONS:
Behavioral: Obesity Prevention Group
  Arms: Obesity Prevention Group
Behavioral: Injury Prevention Group
  Arms: Injury Prevention Group

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial among 468 Non-Hispanic black mothers and their families to test the efficacy of MOTHERS AND OTHERS, a multi-component home visitation program, compared to an attention control (child safety) in promoting appropriate weight gain during infancy.

DETAILED DESCRIPTION:
Mothers and Others: Family-based Obesity Prevention for Infants and Toddlers will be one of the first to meet the unique needs of individual families by delivering anticipatory guidance on infant care, feeding and growth through multiple channels and to multiple caregivers. Primary modes of delivery for the Obesity Prevention Group (experimental arm) will include face-to-face counseling through 8 home visits (1 by a certified Lactation Consultant), 5 health newsletters, and approximately 160 cue-based text messages. The Injury Prevention Group (active comparator) will receive messages on child safety delivered through similar channels. Our main outcome is infant/toddler growth, captured by mean weight-for-length z-scores (WLZ) at 15 months, mean change in WLZ between 0-15 months, and likelihood of overweight (WLZ ≥ 95th percentile) at 15 months. Differences between groups are expected to be achieved through uptake of targeted health behaviors, including a greater likelihood of breastfeeding initiation, exclusivity and duration; after 6 months, higher dietary intakes of whole fruits and vegetables and lower intakes of energy-dense snack foods; age-appropriate durations of infant and toddler sleep; and, lower levels of television and electronic media exposure. We further hypothesize that these targeted health behaviors will be achieved through modifiable risk factors underpinning the intervention, namely more positive breastfeeding attitudes; higher levels of parenting and breastfeeding self-efficacy; higher levels of perceived social support; higher responsive feeding style scores; improved accuracy in perceiving infant/toddler weight status; and, diminished parental perceptions of infant fussiness.

ELIGIBILITY:
Inclusion Criteria:

* Self identifies as non-Hispanic, African-American
* Less than 28 weeks pregnant at time of screening and recruitment
* Expecting a singleton birth
* Maternal age at time of birth will be at 18-39 years
* Lives within specified distance of study site
* Not intending to leave study area before expectant child's 15th month of life
* Agreeable to referring another family member/caregiver to participate in the study

Exclusion Criteria:

* Pre-term birth (<= 36 weeks gestation)
* Less than 18 years at time of delivery
* Delivers infant with a congenital anomaly or medical condition that significantly affects feeding (e.g., cleft lip and/or palate, metabolic disease)
* Delivers multiples
* Newborn nursery, neonatal intensive care unit (NICU), or maternity floor stay for 7 or more days after the delivery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Mean weight-for-length z-score at 15 months of age | 15 months of age
  Anthropometrics measured directly in the home by trained study staff

SECONDARY OUTCOMES:
Proportion of infants ever breastfed and exclusively breastfed at 3 and 6 months of age | 3 and 6 months of age
  Measured using an Infant Diet History questionnaire adapted after the Infant Feeding Practices Study II
Proportion of infants fed complementary foods before 4 or 6 months of age | 4 and 6 months of age
  Measured using an Infant Diet History questionnaire adapted after the Infant Feeding Practices Study II
Infant dietary intake of fruits and vegetables, whole grains, desserts and sweets, and salty snacks at 3, 6, 9, 12 and 18 months of age | 3, 6, 9, 12 and 15 months of age
  Measured at 3, 6, 9 and 12 months using an Infant Diet History questionnaire adapted after the Infant Feeding Practices Study II. Measured at 15 months using the Nutrition Data System for Research (NDSR)
Duration of infant sleep (hours of total daily sleep, hours of nocturnal sleep, and number of night awakenings) at 3, 6, 9, 12 and 18 months of age | 3, 6, 9, 12 and 15 months of age
  Measured using the Brief Infant Sleep Questionnaire (BISQ)
Infant exposure to television and electronic media (number of hours of screen time per day, proportion of infants with a T.V. or other media screen in bedroom) at 3, 6, 9, 12 and 18 months of age | 3, 6, 9, 12 and 15 months of age

OTHER OUTCOMES:
Breastfeeding attitude score at 28 and 37 weeks gestation and at 1, 3, 6, 9 and 12 months of age | 28 and 37 weeks gestation and 1, 3, 6, 9 and 12 months of age
  Measured using the Iowa Infant Feeding Attitude Scale
Breastfeeding self-efficacy score at 1, 3, 6, 9 and 12 months | 1, 3, 6, 9 and 12 months of age
  Measured using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF)
Social support from family score at 1, 3, 6, 9 and 12 months of age | 1, 3, 6, 9 and 12 months of age
  Measured using the Perceived Social Support from Family Scale
Responsive feeding style score at 28 and 37 weeks gestation and 1, 3, 6, 9, 12 and 15 months of age | 28 and 37 weeks gestation and at 1, 3, 6, 9, 12 and 15 months of age
  Measured using the Infant Feeding Styles Questionnaire (IFSQ) (belief items only at 28 and 37 weeks gestation, full scale at all other time points) and the Responsiveness to Child Feeding Cues Scale (RCFCS)at 3, 9 and 15 months.
Perception of infant fussiness (i.e. IBQ-R 'Distress to Limitations' score and 'Activity' score) at 3, 6, 9 and 12 months of age | 3, 6, 9 and 12 months of age
  Measured using the Infant Behavior Questionnaire-Revised (IBQ-R)
Change in weight-for-length z-score between birth to 15 months | Birth to 15 months
  Anthropometrics measured directly in the home by trained study staff
Proportion of infants that are overweight, defined as weight-for-length z-score ≥ 95th percentile, at 15 months | 15 months of age
  Anthropometrics measured directly in the home by trained study staff

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Bentley, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Heather Wasser, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- Center for Women's Health Research, University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Wasser HM, Thompson AL, Suchindran CM, Goldman BD, Hodges EA, Heinig MJ, Bentley ME. Home-based intervention for non-Hispanic black families finds no significant difference in infant size or growth: results from the Mothers & Others randomized controlled trial. BMC Pediatr. 2020 Aug 18;20(1):385. doi: 10.1186/s12887-020-02273-9. PMID 32811460
- [Derived] Wasser HM, Thompson AL, Suchindran CM, Hodges EA, Goldman BD, Perrin EM, Faith MS, Bulik CM, Heinig MJ, Bentley ME. Family-based obesity prevention for infants: Design of the "Mothers & Others" randomized trial. Contemp Clin Trials. 2017 Sep;60:24-33. doi: 10.1016/j.cct.2017.06.002. Epub 2017 Jun 21. PMID 28600160